CLINICAL TRIAL: NCT00739596
Title: An 8 Week Prospective, Multicenter, Randomized, Double-Blind, Active Control, Parallel Group Study to Evaluate the Efficacy and Safety of Aliskiren HCTZ Versus Amlodipine in African American Patients With Stage 2 Hypertension
Brief Title: Blood Pressure Lowering of Aliskiren Hydrochlorothiazide (HCTZ) Versus Amlodipine in Stage 2 Hypertension in African Americans
Acronym: ATLAAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPP100AUS03
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2011-02

CONDITIONS: Hypertension
Keywords: Hypertension; African American; aliskiren; hydrochlorothiazide; systolic blood pressure; diastolic blood pressure; amlodipine; stage 2
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren Hydrochlorothiazide (HCTZ) (Experimental)
  Interventions: Drug: Aliskiren Hydrochlorothiazide (HCTZ): 8 weeks
- Amlodipine (Active Comparator)
  Interventions: Drug: Amlodipine: 8 weeks

INTERVENTIONS:
Drug: Aliskiren Hydrochlorothiazide (HCTZ): 8 weeks — Aliskiren HCTZ (150/12.5 mg) for 1 week followed by forced titration to Aliskiren HCTZ (300/25 mg) for remaining 7 weeks
  Arms: Aliskiren Hydrochlorothiazide (HCTZ)
Drug: Amlodipine: 8 weeks — Amlodipine 5 mg for 1 week followed by forced titration to Amlodipine 10 mg for remaining 7 weeks
  Arms: Amlodipine

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of a fixed dose combination of aliskiren HCTZ versus amlodipine in African American patients with Stage 2 hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible and able to participate in the study, and who give written informed consent before any assessment is performed.
* Men or women 18 years and older of African American background; self identified
* Patients with stage 2 hypertension. Patients must have a MSSBP ≥ 160 mmHg and < 200 mmHg at Visit 5 (randomization)

Exclusion Criteria:

* Office blood pressure measured by cuff (MSSBP ≥ 200 mmHg and/or MSDBP ≥ 110 mmHg) at any visit.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives whichever is longer.
* History of hypersensitivity to any of the study drugs or to drugs belonging to the same therapeutic class (CCBs or thiazide diuretics) as the study drugs.
* Long QT syndrome or QTc > 450 msec for males and > 470 msec for females at screening.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant. including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method.

  1. Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent. Reliable contraception should be maintained throughout the study and for 7 days after study drug discontinuation.
  2. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL [and estradiol < 20 pg/mL] or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* History or evidence of a secondary form of hypertension.
* Known Keith-Wagener Grade III or IV hypertensive retinopathy.
* History of cerebrovascular accident, transient ischemic cerebral attack (TIA), heart failure (NYHA Class II-IV), myocardial infarction, coronary bypass surgery, or any percutaneous coronary intervention (PCI) in the last 12 months.
* Current angina pectoris requiring pharmacological therapy.
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Sites in USA, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Ferdinand KC, Pool J, Weitzman R, Purkayastha D, Townsend R. Peripheral and central blood pressure responses of combination aliskiren/hydrochlorothiazide and amlodipine monotherapy in African American patients with stage 2 hypertension: the ATLAAST trial. J Clin Hypertens (Greenwich). 2011 May;13(5):366-75. doi: 10.1111/j.1751-7176.2010.00416.x. Epub 2011 Jan 18. PMID 21545398

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren Hydrochlorothiazide (HCTZ): Aliskiren HCTZ (150/12.5 mg) for 1 week followed by forced titration to Aliskiren HCTZ (300/25 mg) for remaining 7 weeks
- Amlodipine: Amlodipine 5 mg for 1 week followed by forced titration to Amlodipine 10 mg for remaining 7 weeks
Period: Overall Study
Arm/Group | Aliskiren Hydrochlorothiazide (HCTZ) | Amlodipine
Started | 166 | 166
Completed | 141 | 149
Not Completed | 25 | 17
Not completed — Adverse Event | 12 | 6
Not completed — Unsatisfactory Therapeutic Effect | 4 | 0
Not completed — Patient Withdrew Consent | 8 | 8
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Deviation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Aliskiren HCTZ: Aliskiren HCTZ (150/12.5 mg) for 1 week followed by forced titration to Aliskiren HCTZ (300/25 mg) for remaining 7 weeks
- Total: Total of all reporting groups
Arm/Group | Aliskiren HCTZ | Amlodipine | Total
Number analyzed (Participants) | 166 | 166 | 332
Age, Customized [Number; unit: participants]
  < 65 years | 141 | 143 | 284
  ≥ 65 years | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (11.27) | 53.1 (11.56) | 52.6 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 91 | 176
  Male | 81 | 75 | 156

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (MSSBP) After 8 Weeks of Treatment
Description: To assess the change from baseline in MSSBP after 8 weeks of treatment with an aliskiren HCTZ-based treatment regimen (aliskiren HCTZ 150/12.5 mg, 300/25 mg) versus an amlodipine-based treatment regimen (amlodipine 5 mg, 10 mg) in African American patients with stage 2 hypertension.
Time Frame: Baseline and 8 weeks
Population: The intent-to-treat (ITT) population consisted of all randomized patients who received at least one dose of study medication and had at least one valid post-baseline assessment of the primary efficacy variable. Last observation carried forward (LOCF) method was used for replacing missing values with post-baseline assessments.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren HCTZ | Amlodipine
Number analyzed (Participants) | 162 | 162
mm Hg
  Baseline | 168.2 (8.49) | 168.1 (7.99)
  Week 8 | 138.8 (18.21) | 139.1 (14.45)
  Change from baseline to Week 8 | -29.4 (17.95) | -29.0 (13.17)

2. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (MSDBP) After 8 Weeks of Treatment
Description: To assess the change from baseline in mean sitting diastolic blood pressure (MSDBP) after 8 weeks of treatment with an aliskiren HCTZ-based treatment regimen (aliskiren HCTZ 150/12.5 mg, 300/25 mg) versus an amlodipine-based treatment regimen (amlodipine 5 mg, 10 mg) in African American patients with stage 2 hypertension.
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren HCTZ | Amlodipine
Number analyzed (Participants) | 162 | 162
mm Hg
  Baseline | 96.0 (9.76) | 95.0 (8.86)
  Week 8 | 86.0 (12.02) | 84.0 (9.72)
  Change from Baseline to Week 8 | -10.0 (11.08) | -11.0 (9.81)

3. Secondary Outcome: Change in Mean Sitting Pulse Pressure (MSPP) After 8 Weeks of Treatment
Description: To compare the change from baseline in mean sitting pulse pressure (MSPP) after 8 weeks of treatment with an aliskiren HCTZ-based treatment regimen (aliskiren HCTZ 150/12.5 mg, 300/25 mg) versus an amlodipine-based treatment regimen (amlodipine 5 mg, 10 mg) in African American patients with stage 2 hypertension.
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren HCTZ | Amlodipine
Number analyzed (Participants) | 162 | 162
mm Hg
  Baseline | 72.2 (12.10) | 73.1 (11.59)
  Week 8 | 52.7 (14.91) | 55.1 (12.13)
  Change from Baseline to Week 8 | -19.4 (13.73) | -18.0 (11.20)

4. Secondary Outcome: Percentage of Responders After 8 Weeks of Treatment.
Description: To compare the percentage of responders after 8 weeks of treatment with an aliskiren HCTZ based treatment regimen (aliskiren HCTZ 150/12.5 mg, 300/25 mg) versus an amlodipine-based treatment regimen (amlodipine 5 mg, 10 mg) in African American patients with stage 2 hypertension: [ Responders were defined as patients with MSSBP < 140 mm Hg or a decrease from baseline ≥ 20 mm Hg at 1st response. A response was counted when a patient first achieved MSSBP < 140 mm Hg or a decrease from baseline ≥ 20 mm Hg.]
Time Frame: 8 weeks
Population: The intent-to-treat (ITT) population consisted of all randomized patients who received at least one dose of study medication and had at least one valid post-baseline assessment of the primary efficacy variable.
Measure: Number; unit: Cumulative percentage of responders
Arm/Group | Aliskiren HCTZ | Amlodipine
Number analyzed (Participants) | 162 | 162
Cumulative percentage of responders | 84.6 [-13.92 to 1.58] | 90.7 [13.92 to 1.58]

5. Secondary Outcome: Percentage of Participants Achieving BP Control After 8 Weeks of Treatment
Description: To compare the percentage of patients achieving BP control (<140/90 mm Hg) after 8 weeks of treatment with an aliskiren HCTZ-based treatment regimen (aliskiren HCTZ 150/12.5 mg, 300/25 mg) versus an amlodipine-based treatment regimen (amlodipine 5 mg, 10 mg) in African American patients with stage 2 hypertension.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Number; unit: Cumulative percentage of participants
Arm/Group | Aliskiren HCTZ | Amlodipine
Number analyzed (Participants) | 162 | 162
Cumulative percentage of participants | 63.6 [-9.90 to 12.37] | 62.3 [-9.90 to 12.37]

ADVERSE EVENTS:
Time Frame: 8 Weeks
Arm/Group | Aliskiren HCTZ | Amlodipine
Serious Adverse Events (participants affected / at risk) | 5/166 | 3/166
Other Adverse Events (participants affected / at risk) | 0/166 | 0/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren HCTZ (N=166) | Amlodipine (N=166)
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Encephalitis herpes (Infections and infestations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.